CLINICAL TRIAL: NCT01138540
Title: Prospective, Randomized, Multi-Center Trial of Lateral Trendelenburg Versus Semi-Recumbent Body Position in Mechanically Ventilated Patients For The Prevention of Ventilator-Associated Pneumonia
Brief Title: The Gravity-VAP (Ventilator-Associated Pneumonia) Trial
Acronym: Gravity-VAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Steering Committee accepted DSMB advise to terminate the study after review of data analysis at second interim analysis
Sponsor: Policlinico Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Ospedale Nuovo del Mugello (Unknown); Ospedale San Donato (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); Ospedale S. Giovanni Bosco (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda Ospedaliero-Universitaria di Modena (Other); Ospedale Città di Sesto San Giovanni (Unknown); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Goethe University (Other); Clinical Hospital Centre Zagreb (Other); Santa Chiara Hospital (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Mauro Panigada, MD, MD, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gravity-VAP Trial
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Ventilator Associated Pneumonia
Keywords: VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semirecumbent position (Active Comparator): Semirecumbent position of patients on mechanical ventilation in the bed of the ICU
  Interventions: Other: lateral-Trendelenburg position
- lateral-Trendelenburg position (Experimental): lateral-Trendelenburg position of patients on mechanical ventilation in the bed of the ICU
  Interventions: Other: lateral-Trendelenburg position

INTERVENTIONS:
Other: lateral-Trendelenburg position — lateral-Trendelenburg position of patients laying in the bed of the ICU, keeping trachea and tracheal tube horizontal, compared to the standard treatment (semirecumbent position) for the prevention of VAP

SUMMARY:
This study is planned to compare, in patients sedated, intubated and mechanically ventilated, the efficacy and safety of the Lateral Trendelenburg position in comparison to the Semirecumbent Position to prevent incidence of ventilator-associated pneumonia (VAP).

DETAILED DESCRIPTION:
This study is planned to compare, in patients sedated, intubated or tracheostomized and mechanically ventilated, the efficacy and safety of two body positions in reducing incidence of ventilator-associated pneumonia. The semi-recumbent position prevents gastro-oropharyngeal aspiration of bacteria laden gastric contents and the "gastro-pulmonary" route of colonization. The lateral-Trendelenburg position aims to promote outward drainage of bacteria-laden oropharyngeal secretion, while avoiding bacterial translocation from the oropharynx into the lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients expected to be oro-tracheally intubated for at least 48 hours or longer
3. Enrollment time window within 12 hours following intubation

Exclusion Criteria:

1. Current and past participation in an other intervention trial conflicting with the present study
2. Previous endotracheal intubation longer than 12 hours during the previous 30 days
3. Patients with documented bronchiectasis
4. Cystic fibrosis
5. Witnessed pulmonary aspiration either prior or at intubation
6. Patients with increased intracranial pressure, brain edema; or medical conditions that can worsen with increase in intracranial pressure
7. Patients with significant heart failure and activity impairment (Class III-IV of the New York Heart Association (NYHA)
8. Spinal cord injury
9. BMI > 35, or weight above 300 pound
10. Grade IV Intra-abdominal pressure: IAP > 25 mmHg or abdominal compartment syndrome , defined as a sustained IAP > 20 mmHg that is associated with new organ dysfunction / failure
11. Pregnancy
12. Orthopedic problems that will not allow the patient to be kept in one of the study positions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2010-11 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of ventilator-associated pneumonia | 14 days of mechanical ventilation
  incidence of ventilator-associated pneumonia within the first 14 days of intubation, confirmed by quantitative microbiology analysis of either bronchoalveolar lavage (BAL) or mini-BAL fluids or secretions collected through protected specimen brush (PSB)

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 14 days
Duration of intensive care unit stay | days
Duration of hospital stay | days
Safety of the Semi-Recumbent and Lateral-Trendelenburg position | 14 days
Use of Sedatives | 14 days
Use of Antimicrobials | 14 days
ICU mortality | 28 days
Hospital mortality | 28 days
28 Days mortality | 28 days
Assessment of nursing-related issues in the lateral-Trendelenburg position | 14 days

CONTACTS AND LOCATIONS:
Locations (2):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Mi, Italy
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Derived] Li Bassi G, Panigada M, Ranzani OT, Zanella A, Berra L, Cressoni M, Parrini V, Kandil H, Salati G, Selvaggi P, Amatu A, Sanz-Moncosi M, Biagioni E, Tagliaferri F, Furia M, Mercurio G, Costa A, Manca T, Lindau S, Babel J, Cavana M, Chiurazzi C, Marti JD, Consonni D, Gattinoni L, Pesenti A, Wiener-Kronish J, Bruschi C, Ballotta A, Salsi P, Livigni S, Iotti G, Fernandez J, Girardis M, Barbagallo M, Moise G, Antonelli M, Caspani ML, Vezzani A, Meybohm P, Gasparovic V, Geat E, Amato M, Niederman M, Kolobow T, Torres A; Gravity-VAP Network. Randomized, multicenter trial of lateral Trendelenburg versus semirecumbent body position for the prevention of ventilator-associated pneumonia. Intensive Care Med. 2017 Nov;43(11):1572-1584. doi: 10.1007/s00134-017-4858-1. Epub 2017 Jun 20. PMID 29149418